CLINICAL TRIAL: NCT05228990
Title: Clinical Study on Efficacy and Safety of Warm Acupuncture in Treatment of Cold-sensitive Fibromyalgia Syndrome
Brief Title: Pilot Study of Warm Acupuncture in Treatment of Cold-sensitive Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Juan Jiao, Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CI2021A015
Record Dates: First submitted 2022-01-25; First posted 2022-02-08 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; cold-sensitive; needle warming moxibustion; randomized controlled trial; warm acupunctrue
MeSH Terms: conditions — Fibromyalgia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Warm acupuncture - observation group (Experimental): Sequence A: Participants will receive warm acupuncture for 20 minutes twice a week for eight weeks.
  Sequence B: Patients will be observed without any intervention for eight weeks.
  Interventions: Device: warm acupunctrue
- Observation - warm acupuncture group (Experimental): Sequence A: Patients will be observed without any intervention for eight weeks. Sequence B: Participants will receive warm acupuncture for 20 minutes twice a week for eight weeks.
  Interventions: Device: warm acupunctrue

INTERVENTIONS:
Device: warm acupunctrue — The sterile acupuncture needle (0.3mm×40mm) is taken, and the acupuncture needle is vertically inserted into the corresponding depth of the acupoint. After the needle is transported to "get qi", moxibustion will be added at acupoints. The moxibustion distance is about 3cm from the skin, and the local temperature is warm and the patient felt comfortable with the skin. Replace it after burning out. During the acupuncture treatment, in order to avoid burns, it is necessary to strictly control the distance between moxibustion and skin. In the supine position, cardboard should be placed between moxibustion and skin to prevent burns, and ashes should be removed after moxibustion is completely burned. The needle is left for 20 minutes.
  Other Names: warm needling method; needle warming moxibustion; acupuncture with warmed needle

SUMMARY:
Non-pharmaceutical therapies, such as acupuncture, hydrotherapy, and meditative exercises (such as Qigong (including Tai Chi and Ba-Duan-Jin), have been shown to reduce pain and improve physical function. The management recommendations of fibromyalgia issued by the European Union, Canada, Germany and Israel have all affirmed the "first-line" role of Non-pharmaceutical therapy. Because of its good efficacy and safety, acupuncture therapy has been recommended in the management guidelines and has broad application prospects. Warm acupuncture is a therapy combining acupuncture and moxibustion, which is widely used in the treatment of various painful diseases in China, especially for cold-sensitive patients . This study aims to observe the safety and effectiveness of warm acupuncture in the treatment of cold-sensitive fibromyalgia patients, in order to provide a more alternative non-drug therapy for this particular type of patients with fibromyalgia .

ELIGIBILITY:
Inclusion Criteria:

1. Meet the 1990 American College of Rheumatology (ACR) Research Classification Criteria for fibromyalgia;
2. Be over 18 years of age;
3. The type and dose of drugs used for fibromyalgia should be stable for at least 2 weeks;
4. The VAS score of item 10 (sensitivity to cold) in FIQR scale ≧4 points;
5. Sign informed consent.

Exclusion Criteria:

1. Patients suffering from systemic or local acute infectious diseases;
2. Patients with severe visceral diseases or physical weakness who cannot tolerate acupuncture treatment;
3. Pregnant women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The change of the VAS score for item 10 (susceptibility to cold) of the modified fibromyalgia Impact Questionnaire from baseline. | Baseline, week4, week8, week12, week16
  range from 0 to 10 cm with higher score indicating more sensitive to cold.

SECONDARY OUTCOMES:
The change of the revised Fibromyalgia Impact Questionnaire (FIQR) from baseline | Baseline, week4, week8, week12, week16
  A self-administered questionnaire with 10 subscales, measuring fibromyalgia symptoms and function domains. FIQR total score ranges from 0 to 100, with higher scores indicating more severe symptoms.
The change of the Visual Analogue Scale (VAS) for pain from baseline. | Baseline, week4, week8, week12, week16
  Pain VAS, range, 0 to 10 cm, where higher scores indicated the perceived pain to be more severe.
The change of the Multidimensional Fatigue Inventory-20 (MFI-20) from baseline. | Baseline, week4, week8, week12, week16
  The Multidimensional Fatigue Inventory-20 (MFI-20) measures fatigue severity. The MFI-20 total score ranges from 0 to 80, with higher scores indicate more severe fatigue.
The change of the Perceived Stress Scale (PSS) from baseline. | Baseline, week4, week8, week12, week16
  The Perceived Stress Scale (PSS) is for measuring the perception of stress and The Perceived Stress Scale (PSS) is for measuring the perception of stress and current levels of experienced stress. Scores range from 0 to 56, with higher total score indicating a greater degree of symptom severity
The change of the Hamilton Anxiety Scale（HAMA） from baseline. | Baseline, week4, week8, week12, week16
  he Hamilton Anxiety Scale is used to assess the severity of anxiety symptoms and consists of 14 items, with higher scores indicating greater anxiety
The change of the Beck II Depression Inventory (BDI) from baseline. | Baseline, week4, week8, week12, week16
  The Beck II Depression Inventory (BDI) assesses the severity of depressive symptoms. Scores range from 0 to 39, with higher scores indicate a greater degree of depression severity.
The change of the Short Form-36 Health Status Questionnaire (SF-36) from baseline. | Baseline, week4, week8, week12, week16
  The Short Form-36 Health Status Questionnaire (SF-36), which measured health-related quality of life (range, 0 to 100, with higher scores indicating better perceived health status
The change of the Minimum Mental State Examination(MMSE) from baseline. | Baseline, week4, week8, week12, week16
  The Minimum Mental State Examination(MMSE) scores range from 0 to 30, with higher scores indicating better cognitive function
The change of the Pittsburgh Sleep Quality Index (PSQI) from baseline. | Baseline, week4, week8, week12, week16
  Scores on the Pittsburgh Sleep Quality Index (PSQI) range from 0 to 21, with higher scores indicating worse sleep quality.
Global Impression of Change (PGIC) questionnaire evaluated at week 16. | week16
  A questionnaire determine any change in overall symptom status from the beginning of the study to its conclusion (score range, 1 [very much improved] to 7 [very much worse).

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No